CLINICAL TRIAL: NCT04542369
Title: Neoadjuvant PD-1 Inhibitor (Tislelizumab) Plus Chemotherapy in Patients With Limited-stage Small-cell Lung Cancer: an Open-lable, Single-arm, Phase 2 Trial
Brief Title: Pilot Study of PD-1inhibitor (Tislelizumab) Plus Chemotherapy as Neoadjuvant Therapy for Limited-Stage Small-Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of science and education department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-006 (FK-LYIB-001)
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — tislelizumab; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LS-SCLC (Experimental): Induction therapy: Tislelizumab 200mg, i.v., q3w, 4 cycles; cisplatin 75mg/m2, d1-3 or carboplatin AUC5, d1+ etoposide 100mg/m2, q3w, 4 cycles.
  Regional therapy: Candidates for complete resection will receive surgery otherwise they will receive radiotherapy.
  Adjuvant therapy: Patients received surgery will receive adjuvant Tislelizumab plus platinum-etoposide therapy for four cycles.
  Interventions: Drug: Tislelizumab (BGB-A317) Plus Chemotherapy (Cisplatin/Carboplatin and Etoposide)

INTERVENTIONS:
Drug: Tislelizumab (BGB-A317) Plus Chemotherapy (Cisplatin/Carboplatin and Etoposide) — Inductive/neoadjuvant therapy: Tislelizumab + EP Maintenance/adjuvant therapy: Tislelizumab + EP

SUMMARY:
This is a phase II, non-randomized, open-label, single-center study to evaluate the efficacy and safety of neoadjuvant PD-1 inhibitor (Tislelizumab) + chemotherapy (cisplatin/carboplatin + etoposide) followed by radical surgery and adjuvant Tislelizumab immunotherapy as first-line treatment in patients limited-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form.
2. Aged 18 ≥ years.
3. Histological or cytological diagnosis of SCLC by needle biopsy, and limited stage (local advanced) confirmed by imageological examinations.
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
5. Life expectancy is at least 12 weeks.
6. At least 1 measurable lesion according to RECIST 1.1.
7. Patients with good function of other main organs (liver, kidney, blood system, etc.):

   * ANC count ≥1.5×10^9/L, platelet count ≥100×10^9/L#hemoglobin

     ≥90 g/L;
   * the international standard ratio of prothrombin time (INR) and prothrombin time (PT) < 1.5 times of upper limit of normal (ULN);
   * partial thromboplastin time (APTT) ≤1.5×ULN;
   * total bilirubin ≤1.5×ULN;
   * alanine aminotransferase (ALT) aspartate aminotransferase (AST) ≤2.5×ULN, or ALT and AST ≤5×ULN in the patients with liver metastatic tumor.
8. No systemic metastasis;
9. Expected to be completely resected;
10. Good cardiopulmonary function and can tolerate surgical treatment;
11. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of Tislelizumab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
12. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of Tislelizumab (whichever is later).

Exclusion Criteria:

1. Participants who have received any systemic anti-cancer treatment for SCLC, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
2. Participants with cancer other than SCLC (excluding cervical carcinoma in situ, cured basal cell carcinoma, bladder epithelial tumor [including TA and tis]) within five years before the start of this study;
3. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
4. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
5. Participants who are allergic to the test drug or any auxiliary materials;
6. Have or currently have interstitial lung disease;
7. Participants with active HIV;
8. Antibiotics were used to treat the infection for 4 weeks prior to the start of the trial;
9. Pregnant or lactating women;
10. Any conditions of malabsorption;
11. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
12. Other factors that researchers think it is not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety: frequency of severe adverse events | up to 18 months
  The frequency of severe adverse events from the participants enrolling to 90 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 60 months
  It refers to the time from the first administration of Tislelizumab in this study to the disease progression or death (including any cause of death in the case of no progression) as recorded in CRF, regardless of whether the patient exits from the treatment or receives other anti-cancer treatment before progression.
Overall survival (OS) | up to 63 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Health related quality of life (HRQol) | up to 12 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.
Major pathologic response (MPR) | up to 5 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.
Objective response rate (ORR) | up to 4 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the inductive/neoadjuvant therapy.
  Only patients with measurable lesions at baseline will be analyzed.
Disease-free survival (DFS) | up to 60 months
  It refers to the time from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published